CLINICAL TRIAL: NCT05402969
Title: Evaluation of Electrode-modiolus Distance and Cochlear Fibrosis Using Depth Sounding and Spectroscopy Tools: Comparison With Postoperative Cone Beam CT
Brief Title: Evaluation of Electrode-modiolus Distance and Cochlear Fibrosis Using Depth Sounding and Spectroscopy Tools
Acronym: TIMAGING
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0666
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Sensorineural Hearing Loss; Fibrosis
Keywords: Cochlear implantation; Cochlear fibrosis; Transimpedance matrix measurement; Cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural; Fibrosis | interventions — Spectrum Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with long-term implantation: Patients undergone CI more than 6 months ago. After the study is presented to the patient and the egligibility criterias are verified, the patient is proposed to sign a consent form (visit 0). Once the consent form is signed, the visit 1 is scheduled (0 to 90 days after the visit 0). During the visit 1 TIM measurements are performed, including depth sounding and spectroscopy, and adversed affects if any are collected.
  Interventions: Procedure: Transimedance Matrix measurements; Procedure: Depth sounding and spectroscopy; Procedure: Cone Beam Computer Tomography
- Recently implanted patients: Patients enrolled at their pre-op appointments (visit 0 - egligibilty criterias are verified and the consent collected). Visit 1 (0 to 90 days after visit 0) is a surgery. TIM measurements, icluding deep sound and spectroscopy, are performed after the CI and all adverse events are noted. CBCT is routinely done the next day after CI. TIM measurements (as well as adverse event collection) are repeated during visits 2, 3, 4, 5 and 6 (appoitments 15 days, 1, 2, 3 and 6 months after the surgery).
  Interventions: Procedure: Transimedance Matrix measurements; Procedure: Depth sounding and spectroscopy; Procedure: Cone Beam Computer Tomography

INTERVENTIONS:
Procedure: Transimedance Matrix measurements — TIM measurements are based on cochlear implant back-telemetry function. Each electrode contact is stimulated in monopolar mode. Transimpedance is represented by the ratio between the voltage measured at each recording electrode and the current injected at the stimulation contact. The result of the measurements is a matrix of 21x21 transimpedances. Stimulation current cannot be perceived by a patient thus making TIM measurements a non-invasive and painless procedure. The test duration is only 2-3 minutes
  Other Names: TIM measurements
Procedure: Depth sounding and spectroscopy — Depth sounding and spectroscopy are based on the matrixes obtained after TIM imaging. Deep sounding measures the capacitances throughout the electrode array whereas spectroscopy determines the phase of every transimpedance value. These tests take 10 to 15 minutes together. The stimulation intensity used by depth sounding technique can be perceived by a patient. If it is considered as unpleasant, the test will be stopped.
Procedure: Cone Beam Computer Tomography — CBCT is a routine postoperative assessment after CI, non-invasive and painless for patients.
  Other Names: CBCT

SUMMARY:
Cochlear fibrosis development can compromise the success and the outcomes of the cochlear implantation (CI) thus affecting the quality of life of the implanted patient. Correlating the results of the Transimpedance Matrix (TIM) measurements to the implant electrode location determined by the Cone Beam Computer Tomography (CBCT), this study aims to identify a range of TIM profiles within the implanted population, certain profiles suggesting the growth of the fibrosis tissue in cochlea

DETAILED DESCRIPTION:
Fibrosis tissue growth after the CI is an inflammatory reaction to a foreign body occurring around the electrode array. It is considered responsible for a larger current diffusion, less precise stimulation of auditory nerve fibres and elevated electrical impedances thus affecting the functioning and the battery life of an implant. Fibrosis has been also proposed as a factor reducing residual hearing. Hence, its early detection and prevention can significantly improve the outcomes of CI.

To date, no reliable technique to visualise cochlear fibrosis in vivo exists. However, the TIM measurement developed by Cochlear® including depth sounding and spectroscopy tools could possibly provide a better "view" of the fibrosis apparition after CI. This approach has been already successfully applied in the University Hospital of Montpellier, France, to the patients-users of the Advanced Bionics cochlear implants.

One of the factors provoking the fibrosis tissue development is an electrode positioning into the scala vestibule (SV) versus scala tympani (ST). CBCT will be used to visualise the electrode location as well as possible damages of the inner ear caused by CI. The imaging data will be then linked to the TIM measurements results.

Potential participants will be recruited from the French population of the Cochlear® implant users either coming for their regular checks-up at the ENT service of the University Hospital of Montpellier and implanted for more than 6 month (time necessary for the fibrosis tissue to develop) or recently implanted at the same hospital.

For the patients with long-term implantation (160 participants planned) the TIM measurements will be performed only once whereas the newly implanted group (20 participants planned) will require these measurements to be repeated several times: on the day of the surgery as well as 15 days, 1 month, 2 months, 3 months and 6 months after it. For the first group the post operational CBCT imaging file will be extracted from the patient medical record; for the second group CBCT will be performed during the surgery.

The main objective of this study is:

For the group with long-term implantation - to show the difference in TIM profiles according to the electrode scala position (ST or SV) determined by CBCT 6 months or more after the implantation For the group with recent implantation - to evaluate the changes in TIM profiles with time according to the electrode scala position (ST or SV) determined by CBCT

The secondary objectives are common for both groups:

* To analyse various patient subgroups defined by the electrode type (Contour Advanced - only for long-term implantation, Slim Straight, Slim Modiolar) and the inner ear access (round window, enlarged round window or cochleostomy)
* To identify the TIM profile threshold values, potential indicators of the cochlear fibrosis apparition, depending on the electrode type
* To evaluate the depth sounding tool accuracy for the measurement of the distance between the electrode and the spiral ganglion in comparison to CBCT depending on the type of the electrode array.
* To evaluate the spectroscopy tool accuracy for fibrosis detection in specific cochlear areas (around electrodes dislocated to SV or basal electrodes in case of cohleostomy)

ELIGIBILITY:
Inclusion Criteria:

Group with long-term implantation:

* Age18 years or older
* Affiliation to the French social security
* Signed and dated informed consent form
* Users of uni or bilateral cochlear implants for more than 6 months (CI24CA, CI422, CI512, CI522, CI532, CI612; CI622; CI632), in primo-implantation or reimplantation, with more than 18 electrodes active
* Postoperation CBCT imaging results available

Recently-implanted group:

* Age18 years or older
* Affiliation to the French social security
* Signed and dated informed consent form
* Indication for CI622 or CI632 cochlear implants
* Postoperation CBCT imaging results available

Exclusion Criteria:

* Vulnerable individuals (minors, adults protected in accordance to the French Public Health code, patients deprived of liberty by court decision)
* Daily usage of the cochlear implant for less than 4 hours or weekly usage for less than 5 days
* Failure or disfunction of the cochlear implant

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 160 patients undergone CI more than 6 months ago will be enrolled during their routine checks-up at the University Hospital, Montpellier. This group will include 80 individuals with perimodiolar electrode (Contour Advanced or Slim Modiolar) and 80 individuals with lateral electrode (Slim Straight Array). 20 patients scheduled for CI will be enrolled during their pre-op appointment.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2025-01-12 (Estimated)

PRIMARY OUTCOMES:
TIM profiles in patients with long-term implantation | Visit 1 (0 to 90 days after inclusion)
  Comparison of TIM profiles of patients with ST electrode position versus patients with SV electrode dislocateon in the long-term implantation group
TIM profiles time dynamics in the recently implanted patients | Visit 1 - surgery (0 to 90 days after inclusion), visit 3, 4, 5, 6 (1, 2, 3 and 6 months after surgery)
  Assessment of the TIM profile changes with time and depending on electrode scala position in newly-implanted patients

SECONDARY OUTCOMES:
TIM profiles depending on electrode array and inner ear access | Visit 1 (0 to 90 days after inclusion)
  Comparison of the TIM profiles depending on the electrode array type and inner ear access
Depth sounding versus the distance electrode - spiral ganglion | Visit 1 (0 to 90 days after inclusion)
  Correlation of the depth sounding measures with the electrode-spiral ganglion distance assesed through CBCT imaging
Spectroscopy of the specific electrode insertion zones | Visit 1 (0 to 90 days after inclusion)
  Comparison of the spectroscopy measures in the specific zones prone to electrode insertion damages (180° turn and basal part) between groups with ST electrode positioning and SV electrode dislocation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Montpellier, Montpellier, France